CLINICAL TRIAL: NCT07217314
Title: Multi-Channel Spinal Transcutaneous Electrical Pulsed Stimulation System: STEPSS
Brief Title: Testing a Non-Invasive Spinal Stimulation Device
Acronym: STEPSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gail Forrest (Other)
Responsible Party: Sponsor-Investigator, Gail Forrest, Director, Tim and Caroline Reynolds Center for Spinal Stimulation, Kessler Foundation
Organization: Kessler Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-1283-24
Record Dates: First submitted 2025-09-08; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Participants (Experimental)
  Interventions: Device: Spinal Stimulation

INTERVENTIONS:
Device: Spinal Stimulation — Participants will lay on their back and have small electrodes placed on the center of their backs and several leg muscles. The back electrodes, connected to a battery-operated unit, will send an electrical current to the spine. The leg electrodes will record muscle activity. This will take approximately 2 hours to complete on each day. The 2 hours includes set-up/placement of the electrodes, 4 trials of stimulation with breaks, and removal of electrodes after testing.

SUMMARY:
The purpose of this study is to compare an updated spinal stimulation device with the spinal stimulation device that is currently used. Spinal stimulation is often used in studies aimed at assisting individuals with a spinal cord injury. This device was updated to improve upon limitations in the currently used device.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Proficient in English
* Available for the testing session
* Able to give informed consent
* Able to tolerate spinal stimulation

Exclusion Criteria:

* Pregnant (female only).
* Untreated severe and persistent problems regulating blood pressure, heart rate, or other automatic functions.
* Any past or present injury or disease to the nervous system
* Heart or lung disease that may interfere with stimulation
* A skin condition in any area that may affect the ability to receive stimulation
* Taking any medication that may affect the ability to receive spinal stimulation
* Ongoing drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Leg EMG activity during STEPPS spinal stimulations | up to 6 weeks
  Participants will have electrodes connected to the STEPPS stimulator, placed over spinal site locations (T10/11 & T11/12). These electrodes will send an electrical current to their spine while laying on their back. Additional electrodes will be placed over right leg muscles to measure leg EMG muscle activation during the spinal stimulation. Four trials of stimulation with EMG recording will be given over the course of 2 hours each visit for 3 visits.
  Mean/standard deviation curves and correlation coefficients for right leg muscle activation will be calculated to compare curves for NRT (pre-existing data) and STEPSS stimulators.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States